CLINICAL TRIAL: NCT03358771
Title: Effectiveness and Cost-effectiveness of a COPD Discharge Bundle Delivered Alone or Enhanced Through a Care Coordinator
Brief Title: COPD Discharge Bundle Delivered Alone or Enhanced Through a Care Coordinator
Acronym: PRIHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); Alberta Health services (Other); Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Michael Stickland, Professor, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Pro00065003
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; AECOPD; Discharge care bundle; Patient Care Bundles
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): During the initial stepped wedge phase, all sites will receive usual care. There is currently no standardized discharge care bundle for COPD in Alberta. Some electronic patient information sheets do exist; however, their content is general and use is limited. It is expected that a vast majority of patients will transition to the community on a sub-optimal medication regimen, with limited referral to additional outpatient programs and no formal follow-up organized with a primary care provider (e.g., "F/U prn" or "F/U with Fam MD").
- COPD discharge care bundle (Active Comparator): COPD discharge care bundle:
  1. Ensure patient has demonstrated adequate inhaler technique
  2. Send discharge summary to family physician office and arrange follow-up
  3. Optimize and reconcile prescription of respiratory medications
  4. Provide a written discharge management plan, and assess patient's and care giver's comprehension of discharge instructions
  5. Refer to pulmonary rehabilitation
  6. Screen for frailty and comorbid condition(s)
  7. Assess smoking status, provide counseling and refer to smoking cessation program, where appropriate
  Interventions: Other: COPD discharge care bundle
- COPD discharge care bundle & coordinator (Experimental): COPD discharge care bundle as listed for active comparator arm enhanced with care coordinator support.
  Interventions: Other: COPD discharge care bundle & coordinator

INTERVENTIONS:
Other: COPD discharge care bundle — As a part of RHSCN quality improvement initiative, the elements of the COPD discharge bundle were integrated into a standardized COPD admission order set and are being implemented province-wide. The discharging physician/team will complete the COPD bundle (with reminders facilitated by clinical decision support tools) prior to patient discharge. A copy of the bundle is retained in the patient's medical record, and another copy is sent to the patient's primary care provider detailing the components of the bundle that were completed prior to discharge, and those still needing to be addressed. The patient will also receive a patient-focused discharge checklist detailing discharge bundle items
  Arms: COPD discharge care bundle
Other: COPD discharge care bundle & coordinator — The coordinator will be health professional associated with a Primary Care Network, ED or AHS with access to patient information. Patients will be informed that care coordinator may contact them for follow up after discharge. At 48-72 hours after hospital/ED discharge and then at intervals to be determined, the care coordinator will contact the patient by phone. The care coordinator will identify specific needs or problems that patient may have encountered after discharge, which could potentially affect the successful transition from acute to community care setting. Specifically, the care coordinator will seek information on any follow up with family doctor visit, pulmonary rehabilitation and smoking cessation referrals
  Arms: COPD discharge care bundle & coordinator

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common, chronic progressive lung disease that is characterized by shortness of breath, activity limitation, and a predisposition to flare-ups resulting in frequent emergency department (ED) visits and hospitalizations. COPD flare-ups increase risks of disease progression and mortality and account for the greatest proportion of preventable hospitalizations among major chronic diseases.

Evidence show that timely integrated disease management can prevent future COPD flare-ups and readmissions, but recent data indicate that appropriate follow-up after a COPD hospitalization is limited. To reduce this care gap, the investigators developed a discharge care bundle to help a patient that are being discharged from hospital or ED after COPD flare-up transition to community care.

The aim of this study is to assess how effective and cost-effective is such bundle delivered alone or supported by the dedicated care manager. The investigators will be assessing reduction of ED and hospital readmission.

DETAILED DESCRIPTION:
Introduction/Significance

Chronic obstructive pulmonary disease (COPD) is a common, chronic progressive lung disease that is characterized by shortness of breath, activity limitation, and a predisposition to acute exacerbations resulting in frequent emergency department (ED) visits and hospitalizations. COPD exacerbations account for the greatest proportion of preventable hospitalizations among major chronic diseases. In Alberta, a recent report from the COPD Working Group of the Respiratory Health Strategic Clinical Network (RHSCN) found that, with an average length of stay of 12.9 days, COPD hospitalizations result in an estimated total inpatient cost of $112 million annually. In addition to increasing the risk of disease progression and mortality, COPD exacerbations are a major risk factor for subsequent COPD exacerbations, resulting in additional ED visits and hospitalizations. Approximately 35% of COPD patients who are discharged from the ED have a subsequent revisit within 30 days of initial ED discharge. National data indicate that 18% of hospitalized COPD patients are readmitted within one year after the index hospitalization while 14% are admitted twice within the year. Analysis of Alberta Health Services (AHS) administrative data shows that the 30-day hospital readmission rates for COPD in Alberta during 2012 (18.8%) and 2013 (19.5%) were well above the national 30-day readmission rate for all hospital admissions (8.4%).

The Canadian Thoracic Society (CTS) has developed evidence-based management guidelines for optimizing COPD care and preventing exacerbations and has recommended that COPD patients should be seen by their primary care provider within 14 days following an exacerbation. Further, the Global Initiative for Obstructive Lung Disease has proposed a list of items to review with the patient at discharge and recommends follow-up at 4-6 weeks after discharge. Despite evidence from systematic reviews that timely integrated disease management can prevent future COPD exacerbations and readmissions, recent Alberta data indicate that appropriate follow-up after a COPD hospitalization is limited. An audit at the University of Alberta hospital found that only 43% of COPD patients received appropriate medication prescriptions at discharge; only 10% of eligible patients were referred to a rehabilitation program while only 58% of smokers received instructions on smoking cessation interventions. To overcome these care gaps in COPD, previously published work has supported the introduction of clinical bundles and case management for follow-up after discharge, suggesting promising results to reduce readmissions and minimize health care utilization costs. Clinical bundles support the translation of clinical guidelines into local protocols and their subsequent standardization and application to clinical practice, enhance integrated care, and optimize patient outcomes while maximizing clinical efficiency and containing costs.

A recently completed systematic review of the scientific literature on the effectiveness of COPD discharge care bundles showed that COPD discharge care bundles reduced hospital readmission rates (Risk Ratio [RR]=0.8; 95% Confidence Interval [CI] [0.65, 0.99]); they did not, however, significantly reduce long-term mortality (RR=0.74; CI [0.43; 1.28]) nor improved quality of life after acute care discharge (Mean Difference=1.84; CI [-5.23, 5.80])

COPD discharge care bundle

In view of the promising results from systematic reviews that indicate that integrated care bundles can be effective for conditions with relatively predictable trajectories of care such as COPD, the investigators want to assess whether a COPD discharge bundle adapted to local ED and hospital settings is a relevant, feasible and cost-effective alternative within the Alberta health care system, and whether the addition of a care coordinator to the bundle further reduces ED and hospital readmissions while containing health care costs.

To assure that the care bundle is relevant to the local practice and applicable in the Alberta health system, the research team developed a COPD discharge care bundle through an evidence-based consultation-driven process. During this process, the researchers consulted patients and expert clinicians from Alberta and Canada. The development of the bundle has been a part of 3-year PRIHS project titled "Developing and assessing the effectiveness of a post-discharge care pathway to reduce emergency department revisits and hospital re-admission rates for patients with COPD". The process of bundle development involved several steps:

* Systematic review - to identify evidence-based components incorporated in COPD discharge care bundles in the scientific literature;
* 2-step Delphi technique with field experts and patients to reach consensus on the evidence-based individual components of discharge care bundles;
* A face-to-face Consensus Meeting with practitioners and experts from Alberta and to finalize components of the bundle and identify practical issues for bundle implementation;
* Targeted focus groups with patients and health professionals who work within hospitals, emergency units and/or primary care settings to recognize barriers and facilitators for care bundle implementation.

As a result, the investigators developed the COPD discharge care bundle that includes 7 action items (see Table 2). The list constitutes a single intervention (COPD discharge care bundle). The bundle has subsequently been integrated into the new provincial AHS COPD Order Set by the AHS pathway development team. The current study will specifically examine the efficacy of this new discharge care bundle, and whether the addition of a case manager will improve care. Currently, the research team is conducting the needs and readiness assessments within the five hospitals that are part of the project to determine the best implementation strategies.

Study objectives

This study aims to assess the effectiveness and cost-effectiveness of an evidence-based COPD discharge care bundle, delivered alone or facilitated by a dedicated care coordinator, to reduce ED and hospital readmissions, and improve patient-centered and economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of COPD;
* Male or female, 50 years of age and over, admitted to ED or hospital for an exacerbation of COPD. The age limit is imposed to reduce the chances of enrolling patients with asthma.
* Any stage of severity;
* Not being treated previously under the COPD care bundle

Exclusion Criteria:

* Patients with a diagnosis other than COPD will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3710 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
ED revisits | 30 days after discharge
  Number of revisits
Hospital readmissions | 30 days after discharge
  Number of readmissions

SECONDARY OUTCOMES:
ED revisits | 7 days after discharge
  Number of revisits
ED revisits | 90 days after discharge
  Number of revisits
ED revisits | 1 year after discharge
  Number of revisits
Hospital readmission | 7 days after discharge
  Number of readmissions
Hospital readmission | 90 days after discharge
  Number of readmissions
Hospital readmission | 1 year after discharge
  Number of readmissions
Time to first physician visit and total visits | in the first 30 days after discharge
  Number of days
Time to first physician visit and total visits | in the first 90 days after discharge
  Number of days
Mortality | 7 days after discharge
  Number of cases
Mortality | 30 days after discharge
  Number of cases
Mortality | 90 days after discharge
  Number of cases
Mortality | 1 year after discharge
  Number of cases
Patient Experience - Inpatient | 45-60 days after discharge
  For a randomly selected sample of patients, Patient Experience Survey - Inpatient Care
Patient Experience - ED | 45-60 days after discharge
  For a randomly selected sample of patients, Patient Experience Survey - Emergency Department
Economic Evaluation | 1 year after termination of the trial
  Cost per readmission prevented; cost of intervention; cost of healthcare use (MD visits, ED visits, medication use, hospitalizations)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (5):
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Red Deer Regional Hospital Centre, Red Deer, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atwood CE, Bhutani M, Ospina MB, Rowe BH, Leigh R, Deuchar L, Faris P, Michas M, Mrklas KJ, Graham J, Aceron R, Damant R, Green L, Hirani N, Longard K, Meyer V, Mitchell P, Tsai W, Walker B, Stickland MK. Optimizing COPD Acute Care Patient Outcomes Using a Standardized Transition Bundle and Care Coordinator: A Randomized Clinical Trial. Chest. 2022 Aug;162(2):321-330. doi: 10.1016/j.chest.2022.03.047. Epub 2022 Apr 9. PMID 35405112